CLINICAL TRIAL: NCT00063726
Title: An International, Non-Comparative, Open-Label Study of PS-341 Administered to Patients With Multiple Myeloma Who Experienced Relapsed or Progressive Disease After Receiving at Least Four Previous Treatment Regimens or Experienced Progressive Disease After Receiving Dexamethasone in Millennium Protocol M34101-039
Brief Title: A Study of PS-341 Given to Patients With Multiple Myeloma Who Experienced Progressive Disease After Receiving Dexamethasone in M34101-039
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M34101-040; NCT00049478 (obsolete NCT alias)
Record Dates: First submitted 2003-07-02; First posted 2003-07-11 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
The purpose of this study is to allow patients to receive VELCADE™ (bortezomib) for Injection who experienced progressive disease(PD) while receiving high-dose dexamethasone from the M34101-039 study.

DETAILED DESCRIPTION:
The rationale for Amendment 2 is 2-fold. First, it is intended that this study serve as a rollover protocol for patients who experience progressive disease (PD) after receiving the comparator treatment, high-dose dexamethasone, in MPI Study M34101-039, thereby ultimately providing all patients who participate in Study M34101-039 and require treatment for their disease access to VELCADE™ (bortezomib) for Injection, formerly known as MLN341, LDP-341 and PS-341.

ELIGIBILITY:
Inclusion Criteria

* Patient experienced PD, as defined by SWOG+ criteria during or after treatment with high-dose dexamethasone in MPI Study M34101-039, but has not received alternate anti-neoplastic therapy. Intolerance to high-dose dexamethasone therapy as administered in MPI study M34101-039 does not qualify as PD.
* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Female patient is post-menopausal, surgically sterilized, or willing to use acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) from Screening through the End of Treatment visit.
* Male patient agrees to use an acceptable barrier method for contraception from Screening through the End of Treatment visit.
* Patient meets the following pretreatment laboratory criteria at and within 14 days before Baseline (Day 1 of Cycle 1, before study drug administration). (Note that the End of Treatment assessments of MPI study M34101-039 may qualify as the Screening assessments for MPI study M34101-040 if performed within 14 days of the Baseline visit.):
* Platelet count ≥20 X 10E+9/L, with or without transfusion support.
* Hemoglobin ≥7.0 g/dL, with or without transfusion support.
* Absolute neutrophil count (ANC)≥0.5 x 10E+9/L, without growth factor support.
* Serum calcium <14 mg/dL (3.5 mmol/L).
* Aspartate transaminase (AST):≤2.5 x the upper limit of normal (ULN).
* Alanine transaminase (ALT):≤2.5 x the ULN.
* Total bilirubin:≤1.5 x the ULN.
* If calculated or measured creatinine clearance: ≥20 mL/minute, assessments are as specified in the protocol. If calculated or measured creatinine clearance is <20 mL/minute.

Exclusion Criteria

* Patient participated in M34101-039 and did not have confirmed PD. Dexamethasone intolerance does not qualify as PD.
* Patient had PD on the dexamethasone arm of the MPI Study M34101-039, and then received alternate anti-neoplastic therapy.
* Patient has not recovered from dexamethasone-related toxicity experienced during MPI Study M34101-039.
* Patient is known to be human immunodeficiency virus (HIV)-positive.(Patients assessed by the investigator to be at risk for HIV infection should be tested in accordance with local regulations.)
* Patient is known to be hepatitis B surface antigen-positive or has known active hepatitis C infection.(Patients assessed by the investigator to be at risk for hepatitis B or C infection should be tested in accordance with local regulations.)
* Female patient is pregnant or breast-feeding.
* Patient developed a new or experienced worsening of an existing illness during or after completion of Study M34101-039 that, in the investigator's opinion, may put the patient at risk of participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2002-04; Primary Completion 2005-05 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (76):
- United States (39):
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - City of Hope, Duarte, California
  - Scripps Clinic, Green Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Lombardi Cancer Center, Georgetown University Medical Center, Washington D.C., District of Columbia
  - Med Star Institute, Washington D.C., District of Columbia
  - Hematology/Oncology Associates, PA, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University Medical School, Chicago, Illinois
  - Loyola University Medical Center: Cardinal Bernardin Cancer Center, Maywood, Illinois
  - LSU HC, Sheveport, Louisiana
  - Tufts England Medical Center, Boston, Massachusetts
  - Mass General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Center, Boston, Massachusetts
  - Univ. of Michigan Comp. Cancer Center,, Ann Arbor, Michigan
  - VA Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, David Jurist Research Building, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - Weill Medical College of Cornell University, NY Presbyterian Hospital, New York, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester Medical Center, James P. Wilmot Cancer Center, Rochester, New York
  - Charlotte Hematology Oncology Associates, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Trident Palmetto Hematology/Oncology, Charleston, South Carolina
  - Division of Hematology/Stem Cell Transplant, Nashville, Tennessee
  - Texas Oncology at Medical City Dallas Hospital, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Wilhelminenspital Wien, Abt. Fur Med. und Medizinische Onkologie, Vienna, Austria
- Belgium (5):
  - ACZA, Campus Stuivenberg, Antwerp
  - AZ St. Jan, Dept of Haematology, Bruges
  - Institue Jules Bordet, Unite Sterile, Brussels
  - CHU Erasme / ULB University, Brussels
  - C.H. Notre Dame-Reine Fabiola, Department d'Oncologie et Hematolgie, Charleroi
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - London Health Sciences Center, London, Ontario
  - Toronto General Research Institute, Toronto, Ontario
  - McGill University Clinical Research Program, Montreal, Quebec
- France (7):
  - Hospital Claude Huriez, Lille, Cedex
  - Hoptial Hotel Dieu, Paris, Cedex
  - Hopital Purpan, Pavillon Dieulafoy, Service d'Hematologie Clinique, Toulouse, Cedex
  - Hopital de Brabois, Vandœuvre-lès-Nancy, Cedex
  - Centre Hospitalier Lyon Sud, Cedex
  - Hopital Antoine Beclere, Clamart
  - Hospital Saint-Louis, Paris
- Germany (7):
  - Universitatsklinikum Charite Medizinische Klinik und Poliklinik, Berlin
  - Medizinsche Klinik und Poliklinik 1, Rheinische Friedrich-Wilhelms-Universitaet, Bonn
  - University of Erlangen-Nurenberg, Division of Hematology/Oncology, Erlangen
  - Medical University Clinic (Oncology/Haematology), Hamburg
  - Universitatsklinikum Heidelberg, Heidelberg
  - Johannes-Gutenberg-University Medical School, Department of Medicine III, Mainz
  - Uniklinikum Muenster, Medizinische Klinik und Poliklinik A, Münster
- Belfast City Hospital, Haematology Department, Belfast, Ireland
- Hadassah University Hospital, Jerusalem, Israel
- Italy (2):
  - Dipartimento di Biotecnologie Cellulari ed Ematologia, Az. Policlinico Umberto 1, Roma
  - Azienda Ospedaliera, S. Giovanni Battista, Torino
- Erasmus MC, 1a, Daniel Den Hoed, Department of Hematology, Rotterdam, Netherlands
- Spain (2):
  - Hospital Clinico Universitario de Barcelona, Hematologia, Barcelona
  - University Hospital of Salamanca, Hematology Dept, Salamanca
- Huddinge University Hospital M54, Department of Haematology, Stockholm, Sweden
- United Kingdom (5):
  - Adult Leukaemia Unit, Christie Hospital, Withington, Manchester
  - Queen Elizabeth Hospital, Birmingham
  - Leeds General Infirmary, Department of Haematology, Leeds
  - Department of Haematology, ICSM, London
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] van Duin M, Broyl A, de Knegt Y, Goldschmidt H, Richardson PG, Hop WC, van der Holt B, Joseph-Pietras D, Mulligan G, Neuwirth R, Sahota SS, Sonneveld P. Cancer testis antigens in newly diagnosed and relapse multiple myeloma: prognostic markers and potential targets for immunotherapy. Haematologica. 2011 Nov;96(11):1662-9. doi: 10.3324/haematol.2010.037978. Epub 2011 Jul 26. PMID 21791470